CLINICAL TRIAL: NCT02663999
Title: A Two-Period, Randomized, Open-Label, Crossover Pharmacokinetic Study to Assess Dose Proportionality, Safety and Tolerability of Diazepam Nasal Spray in Healthy Adult Volunteers
Brief Title: A Pharmacokinetic Study to Assess Dose Proportionality, Safety and Tolerability of Diazepam Nasal Spray in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DZNS-PK-1034
Record Dates: First submitted 2016-01-22; First posted 2016-01-26 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
Keywords: dose proportionality; diazepam nasal spray
MeSH Terms: interventions — Diazepam; Nasal Sprays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- diazepam nasal spray (AB) (Experimental): Each subject will receive two single doses of investigational product (DL1, DL2) with a 14-day washout between the doses. The order in which the doses are administered will be randomized, with subjects assigned to 1 of 2 treatment sequences: DL1 (A) followed by DL2 (B), or the reverse order (BA).
  Interventions: Drug: diazepam nasal spray
- diazepam nasal spray (BA) (Experimental): Each subject will receive two single doses of investigational product (DL1, DL2) with a 14-day washout between the doses. The order in which the doses are administered will be randomized, with subjects assigned to 1 of 2 treatment sequences: DL1 (A) followed by DL2 (B), or the reverse order (BA).
  Interventions: Drug: diazepam nasal spray

INTERVENTIONS:
Drug: diazepam nasal spray — diazepam nasal spray at two dose levels (DL). One dose of diazepam nasal spray is administered as two intranasal sprays; one in each nostril using a nasal spray device.
  Other Names: PLUMIAZ™ (diazepam) Nasal Spray

SUMMARY:
This is a single-center, two-period, randomized, open-label, crossover pharmacokinetic (PK) study in healthy adult volunteers to evaluate dose proportionality of diazepam nasal spray using two dose levels

ELIGIBILITY:
Inclusion Criteria:

* Screening body weight 88 to 111 kg, inclusive;
* General good health with no clinically significant abnormalities that would affect ability to complete study as determined by medical history, physical examination, visual evaluation of the septum and turbinates to document baseline anatomy, electrocardiogram, clinical laboratory test results;
* Negative drug and alcohol testing;
* Negative pregnancy test for female subjects of childbearing potential.

Exclusion Criteria:

* Subject who is not surgically sterile or female subject who is less than 2 years postmenopausal, and who does not agree to use a highly effective birth control method during the study and up to 3 months after the last dose of investigational product;
* In the judgment of the Investigator, any clinically significant abnormality (such as septal perforations) or illness that would interfere with participation in this study as determined by medical history, physical examination (including visual exam of septum and turbinates), ECG, clinical laboratory results, or other screening safety tests;
* Any other condition and/or situation that causes the investigator to deem a subject unsuitable for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-01; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Maximum measured plasma concentration (Cmax) | within 15 minutes prior to dosing and at specified time points up to 24 hours post-dose
Area under the concentration curve from time 0 to the concentration at 24 hours (AUC0-24) | within 15 minutes prior to dosing and at specified time points up to 24 hours post-dose
Area under the concentration curve from time 0 to infinity (AUCinf) | within 15 minutes prior to dosing and at specified time points up to 24 hours post-dose
Apparent total body clearance of drug from plasma (CL/F) | within 15 minutes prior to dosing and at specified time points up to 24 hours post-dose

SECONDARY OUTCOMES:
Number of patients with adverse events (AEs) including serious AEs | up to 21 days
Change in focused nasal exam | within 30 minutes prior to dosing and at specified time points up to 24 hours post-dose
Taste change questionnaire | from 5 minutes up to 24 hours post-dose
  If patient reports a change in taste associated with diazepam nasal spray, questionnaire to be completed by research staff.

CONTACTS AND LOCATIONS:
Overall Officials: David Squillacote, MD, Study Director — Acorda Therapeutics
Locations (1):
- Site #001, Dallas, Texas, United States